CLINICAL TRIAL: NCT00001165
Title: Evaluation of Chemotherapy With Streptozotocin Combined With 5-Fluorouracil and Adriamycin in Patients With Zollinger-Ellison Syndrome and Metastatic Non-Beta-Islet Cell Neoplasm
Brief Title: Combination Chemotherapy in Patients With Zollinger-Ellison Syndrome and Tumors of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 780133; 78-DK-0133
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-08

CONDITIONS: Islet Cell Adenoma; Neoplasm Metastasis; Zollinger Ellison Syndrome
Keywords: Gastrinoma; Acid Secretion; Toxicity
MeSH Terms: conditions — Adenoma, Islet Cell; Neoplasm Metastasis; Zollinger-Ellison Syndrome; Gastrinoma | interventions — Streptozocin; Fluorouracil; Doxorubicin

INTERVENTIONS:
Drug: combined chemotherapy with streptozotocin, 5-fluorouracil, and doxorubicin

SUMMARY:
Patients with Zollinger-Ellison Syndrome suffer from ulcers of the upper gastrointestinal tract, higher than normal levels of gastric acid, and tumors of the pancreas known as non-beta islet cell tumors.

Prior to the use of drugs to cure the ulcers, patients typically died due to severe ulcers. Because of such effective drugs to treat the ulcers it is more common to see patients dying due to the pancreatic tumors.

The study will observe patients suffering from Zollinger-Ellison Syndrome and non-beta islet cell tumors and determine the effectiveness of combined chemotherapy with streptozotocin, 5-fluorouracil, and doxorubicin.

DETAILED DESCRIPTION:
Heretofore morbidity and risk of death in Zollinger-Ellison syndrome were caused by severe ulcer disease. The advent of specific drugs to cure ulcer disease now extends life until metastases from the non-beta-islet cell tumor cause death. The present study proposes to continue to test the effect of combined chemotherapy with streptozotocin, 5-fluorouracil and doxorubicin in biopsy-proven cases of metastatic non-beta-islet cell tumor in patients with Zollinger-Ellison syndrome. We published our initial experience with this protocol in 1988. An objective response was observed in 40% of patients.

ELIGIBILITY:
INCLUSION CRITERIA

Subjects selected for this study will be patients with Zollinger-Ellison syndrome who are being evaluated under the protocol entitled "Diagnostic Evaluation of Patients with Suspected Abnormalities of Gastric Secretion" (80-DK-0123).

Histologically proven gastrinoma;

Evidence of metastatic disease or locally invasive tumor by angiography, ultrasound, computerized axial tomography, MRI scan or bone scan;

Progression of the tumor during the preceding 6 months.

EXCLUSION CRITERIA

The following pre-existing conditions will exclude patients from the study:

Congestive heart failure;

Proteinuria greater than 1 gram/day;

Serum creatinine greater than 1.5 mg%;

Platelet count less than 100,000/mm3;

White blood count less than 2500/mm3;

Pregnancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 999
Dates: Start 1978-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), Bethesda, Maryland, United States

REFERENCES:
- [Background] Wolfe MM, Jensen RT. Zollinger-Ellison syndrome. Current concepts in diagnosis and management. N Engl J Med. 1987 Nov 5;317(19):1200-9. doi: 10.1056/NEJM198711053171907. PMID 3309661
- [Background] Moertel CG, Lavin PT, Hahn RG. Phase II trial of doxorubicin therapy for advanced islet cell carcinoma. Cancer Treat Rep. 1982 Jul;66(7):1567-9. PMID 6284361
- [Background] Broder LE, Carter SK. Pancreatic islet cell carcinoma. II. Results of therapy with streptozotocin in 52 patients. Ann Intern Med. 1973 Jul;79(1):108-18. doi: 10.7326/0003-4819-79-1-108. No abstract available. PMID 4352784